CLINICAL TRIAL: NCT03043768
Title: Cutaneous Autonomic Pilomotor Testing to Unveil the Role of Neuropathy Progression in Early Parkinson's Disease (CAPTURE PD)
Brief Title: Cutaneous Autonomic Pilomotor Testing to Unveil the Role of Neuropathy Progression in Early Parkinson's Disease
Acronym: CAPTURE-PD
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Prothena Biosciences Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CAPTURE PD,Vs.02.0,06/29/2015
Record Dates: First submitted 2016-12-28; First posted 2017-02-06 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Autonomic; Diagnosis; Pilomotor; Alpha-synuclein; Axon-reflex; Peripheral nerve fibers
MeSH Terms: conditions — Parkinson Disease; Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3mm skin biopsies (punch biopsies)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PD patients: Male and female PD patients (idiopathic parkinsonism, Hoehn and Yahr [H&Y] scores 1-2) aged 35 to 80 years
- Control subjects: Age-and gender matched healthy control subjects

SUMMARY:
In Parkinson's disease (PD), alpha-synuclein accumulation in cutaneous autonomic pilomotor and sudomotor nerve fibers has been linked to autonomic nervous system disturbances even in the early stages of the disease. The investigators recently introduced a non-invasive technique to assess autonomic adrenergic fiber function using the quantitative pilomotor axon-reflex test (QPART). In the present study the investigators aim to assess the association between alpha-synuclein mediated structural autonomic nerve fiber damage and nerve function in PD, elucidate the role of neuropathy progression during the early disease stages, and test reproducibility and external validity of pilomotor function assessment using quantitative pilomotor axon-reflex test (QPART) and sudomotor function via quantitative direct and indirect test of sudomotor function (QDIRT).

A prospective controlled study will be conducted in four sites (Dresden, Germany; Berlin, Germany; Budapest, Hungary; Boston, USA). A total of 52 male and female patients with idiopathic PD (Hoehn&Yahr 1-2) and 52 age- and sex-matched healthy controls will be recruited. Pilomotor function will be evaluated after iontophoresis of phenylephrine on the dorsal forearm to elicit a cutaneous axon-reflex mediated response (goosebumps). Silicone impressions of the stimulated area will be obtained, scanned and quantified for pilomotor muscle impressions by number, impression size and area of axon-reflex pilomotor erection spread. Sudomotor function will be evaluated after axon-reflex stimulation via iontophoresis of acetylcholine on the dorsal forearm. Stained sweat droplets will be captured using repeated digital photography and will be quantified over time for droplet number and axon-reflex spread. Sympathetic skin responses following deep inspiration will be analyzed using skin conductance quantification. Testing and evaluation of autonomic and motor symptoms will be performed at baseline, after 2 weeks, 1 year, 2 years and 3 years. Skin biopsies will be obtained at baseline and after 3 years and will be analyzed for nerve fiber density and alpha-synuclein accumulation.

The investigators expect that this study will unveil whether progression of autonomic nerve dysfunction assessed via pilomotor and sudomotor axon-reflex tests is related to progression of autonomic symptom severity and alpha-synuclein deposition in PD. Additionally, potential applications of the used techniques include interventional studies evaluating disease-modifying approaches and clinical assessment of autonomic dysfunction in patients with PD.

DETAILED DESCRIPTION:
PURPOSE OF THE PROTOCOL With the goal of developing novel endpoints for early stage trials of disease modifying therapies in Parkinson's disease (PD) the objective of this study is to a) assess reproducibility b) external validity and reliability c) to perform a longitudinal assessment of sudomotor (QDIRT) and pilomotor (QPART) responses in early PD patients.

Moreover, this study aims to assess the hypothesis that functional impairment in pilomotor and sudomotor nerve fibers in early PD correlates with a-synuclein deposition mediated structural fiber damage and may therefore constitute a potential non- invasive biomarker for autonomic involvement in PD.

BACKGROUND In skin biopsy studies of PD, alpha-synuclein accumulation in cutaneous autonomic nerve fibers has been linked to autonomic nervous system disturbances even in the early stages of the disease. (1) The investigators recently introduced a non-invasive technique to assess autonomic adrenergic fiber function using the quantitative pilomotor axon-reflex test (QPART). (2)

OBJECTIVES Demonstrating generalizability and reliability of the QPART technique, the anticipated positive results of this protocol might lend support to the utility of QPART as a diagnostic tool. This might be of particular interest in clinical practice as the QPART technique has been shown to assess small fiber function with low variability and comparatively low technical effort whereas vasomotor assessment is limited by high variability and sudomotor assessment requires technical demanding settings. (3) Moreover, the anticipated positive correlation between functional and structural pilomotor nerve fiber impairment might support the capacity of the QPART technique to assess specific fiber damage and thus provide a non-invasive tool to 1.) study pilomotor nerve damage in research studies and 2.) allow for longitudinal clinical assessment in PD patients to monitor disease progression.

ETHICAL STANDARD The study protocol has been approved by the institutional review board of Technische Universität Dresden (IRB study reference: EK349082015) as well as by the institutional review board of each participating site (Berlin accepted the protocol based on Technische Universität Dresden IRB approval; Budapest IRB number: 004513-004/2016/OTIG; Boston IRB number: 2016P000141)

This study will be conducted according to the principles expressed in the Declaration of Helsinki. Written informed consent will be obtained from each study participant. The consent will be reviewed with the subject by one of the study physicians. The subject will sign the informed consent before any procedures pertaining to the study are initiated. A copy of the signed informed consent will be given to the participant and another copy kept on file. Conduction of this study will comply with the GCP (Good Clinical Practice) guidelines.

STUDY PROCEDURES Quantitative Pilomotor Axon-Reflex Test (QPART): Iontophoresis of phenylephrine is used to induce axon-reflex mediated piloerection. A drug delivery capsule electrode (LI-611; Perimed®, Järfälla, Sweden) is affixed on the testing area on the dorsal forearm. The inner chamber of this capsule, open to the skin surface, is filled with 0.4ml of 1 % phenylephrine solution. The drug delivery electrode is then connected to the iontophoresis stimulation box (Phoresor II-Auto-PM850; IOMED Inc., Salt Lake City, USA). Iontophoresis is performed over a 1cm diameter skin region with 0.5mA over 5 minutes. Silicone impressions of piloerection are obtained to create a local topographic map of piloerection. A silicone based two-phase material with high liquidity (Honigum Light, DMG, Hamburg, Germany) is placed over the skin for 10 seconds. The silicone cures for 5 minutes, has toner applied to mark the pilomotor impressions, excess toner is wiped free and the silicone is scanned to capture the image digitally. Silicone impressions of erect hair follicles are quantified by number and area and spatial spread. A high resolution scanner (Fuel 3D® Technologies Limited, Chinnor, United Kingdom) connected to a personal computer equipped with image analyzing software (Fuel3D® Studio Starter; Fuel 3D® Technologies Limited, Chinnor, United Kingdom) is used to quantify additionally the goosebump reaction.

Sympathetic Skin Response (SSR): The skin conductance level (SCL) is measured in µSievert (µS) from two medial phalanges (index and third finger) with a Powerlab® polygraph (AD Instruments, Bella Vista, Australia). The maximum increase in amplitude following sudden deep respiration (Sympathetic Skin Response; SSR) is calculated to quantify the functional reactivity of sweat glands as previously described. (4)

Quantitative Direct and Indirect Test of Sudomotor Function (QDIRT): Axon-reflex mediated sweating is measured after iontophoresis of 10% acetylcholine by drying the stimulated region on the volar aspect of the forearm and dusting with indicator dye (povidone-iodine and cornstarch) followed by repeated digital photographs taken every 15 seconds for 7 minutes with a 18 Megapixel camera (EOS 60D; Canon Inc., Tokyo, Japan) with 100-mm macro lens. Images are digitally analyzed for droplet number, size, and axon-reflex spread as previously described. (5)

Evaluation of perceived motor and autonomic symptoms: Progression of motor and autonomic symptoms are assessed through validated symptom scores MDS-UPDRS motor part and SCOPA AUT.

Skin biopsies: a-synuclein/PGP Ratio; Immunhistochemical staining for a-synuclein and intraepidermal nerve fibers will be performed in 3 skin punch biopsies obtained from the QPART testing sites and two control sites (lower legs). Three-millimeter biopsies will be obtained following local anesthesia with 2% lidocaine. Biopsy specimens will be fixed in Zamboni solution for 18 hours and cryoprotected overnight (20% glycerol and 20% 0.4 M Sorensen buffer). Skin blocks are cut using freezing microtome and 20 tissue sections are analyzed. 20 tissue sections will analyzed. Alpha synuclein/intraepidermal nerve fiber density ratios will be calculated.

TIMELINE Subjects will be assessed for eligibility by a listed study physician. At baseline all subjects will undergo medical history, physical examination, QPART, SSR, QDIRT, MDS-UPDRS and SCOPA AUT assessment as described above. These testing procedures will be repeated, after 1-2 weeks, 1 year, 2 years, and 3 years post-baseline. All testing will be performed in a temperature and humidity controlled environment. Only at Dresden-Site subjects will additionally undergo the skin punch biopsy procedure as described above at baseline, after 1 year and after 3 years.

ELIGIBILITY:
INCLUSION CRITERIA

- Male and female PD patients (idiopathic parkinsonism, Hoehn and Yahr [H&Y] scores 1-2) aged 35 to 80 years and age-and gender matched healthy control subjects

EXCLUSION CRITERIA

* any dermatological disorders affecting the cutaneous testing regions
* treatment with tricyclic antidepressants, noradrenergic antidepressants, beta-blockers, alpha-adrenergic agonists or antagonists, cholinergic or anti-cholinergic agents
* known allergy to phenylephrine or acetylcholine
* elevated alcohol consumption (more than 4 alcoholic beverages/week)
* nicotine consumption within the past 5 years
* known disorders affecting autonomic functions (including diabetes, pure autonomic failure, inflammatory demyelinating polyradiculoneuropathies, multiple system atrophy, atypical Parkinson syndromes, body mass index over 25 kg/m2, acute or chronic renal disease, gout, rheumatoid arthritis, Lupus, Sjogren 's syndrome, Triple- A syndrome, autonomic neuropathies not related to PD)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients with early Parkinson's disease, gender matched healthy control subjects
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
QPART Pilomotor Function Parameter - Number of goose bump impressions | 36 months
  Mean difference in number of goose bump impressions compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).
QPART Pilomotor Function Parameter - Mean area of goose bump impressions | 36 months
  Mean area of goose bump impressions compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).
QPART Pilomotor Function Parameter - Spatial spread of axon-reflex pilomotor response | 36 months
  Spatial spread of axon-reflex pilomotor response compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).

SECONDARY OUTCOMES:
Alpha-synuclein Ratio | 36 months
  Intraneural alpha-synuclein deposition normalized to intraepidermal small fiber density. Skin biopsies gained with punch biopsy technique.
Perceived Autonomic Symptoms | 36 months
  Autonomic symptom severity tested via the SCOPA AUT (Assessment of autonomic dysfunction in Parkinson's disease) questionnaire.
Motor Symptom Progression | 36 months
  Motor symptom severity tested via the MDS-UPDRS (revised Parkinson's disease rating scale (UPDRS) test).

OTHER OUTCOMES:
QDIRT Sudomotor Function Parameter - Number of Sweat droplets | 36 months
  Number of sweat droplets in the axon-reflex region compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).
QDIRT Sudomotor Function Parameter - Size of sweat droplets | 36 months
  Size of sweat droplets in the axon-reflex region compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).
QDIRT Sudomotor Function Parameter - Axon-reflex spread of sweat droplets | 36 months
  Axon-reflex spread of sweat droplets in the axon-reflex region compared between Cohort 1 (PD Patients) and Cohort 2 (healthy volunteers).
Sympathetic Skin Response | 36 months
  Skin conductance level in µSievert (µS) obtained in two medial phalanges (index and third finger).

CONTACTS AND LOCATIONS:
Overall Officials: Timo Siepmann, MD, Principal Investigator — Department of Neurology, University Hospital Carl Gustav Carus, Technische Universität Dresden; Ben MW Illigens, MD, Principal Investigator — Center for Autonomic and Peripheral Nerve Disorders, Department of Neurology, Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (4):
- Center for Autonomic and Peripheral Nerve Disorders, Department of Neurology, Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts, United States
- Germany (2):
  - Department of Neurology, University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Saxony
  - Departement of Neurology, Charite University Medicine Berlin, Berlin
- Department of Neurology, Semmelweis University, Budapest, Hungary

REFERENCES:
- [Background] Wang N, Gibbons CH, Lafo J, Freeman R. alpha-Synuclein in cutaneous autonomic nerves. Neurology. 2013 Oct 29;81(18):1604-10. doi: 10.1212/WNL.0b013e3182a9f449. Epub 2013 Oct 2. PMID 24089386
- [Background] Siepmann T, Gibbons CH, Illigens BM, Lafo JA, Brown CM, Freeman R. Quantitative pilomotor axon reflex test: a novel test of pilomotor function. Arch Neurol. 2012 Nov;69(11):1488-92. doi: 10.1001/archneurol.2012.1092. PMID 22868966
- [Background] Freeman R. Autonomic peripheral neuropathy. Lancet. 2005 Apr 2-8;365(9466):1259-70. doi: 10.1016/S0140-6736(05)74815-7. PMID 15811460
- [Background] Hu F, Jin J, Qu Q, Dang J. Sympathetic Skin Response in Amyotrophic Lateral Sclerosis. J Clin Neurophysiol. 2016 Feb;33(1):60-5. doi: 10.1097/WNP.0000000000000226. PMID 26844971
- [Background] Gibbons CH, Illigens BM, Centi J, Freeman R. QDIRT: quantitative direct and indirect test of sudomotor function. Neurology. 2008 Jun 10;70(24):2299-304. doi: 10.1212/01.wnl.0000314646.49565.c0. PMID 18541883
- [Derived] Siepmann T, Arndt M, Sedghi A, Szatmari S Jr, Horvath T, Takats A, Bereczki D, Moskopp ML, Buchmann S, Skowronek C, Zago W, Woranush W, Lapusca R, Weidemann ML, Gibbons CH, Freeman R, Reichmann H, Puetz V, Barlinn K, Pinter A, Illigens BM. Two-Year observational study of autonomic skin function in patients with Parkinson's disease compared to healthy individuals. Eur J Neurol. 2023 May;30(5):1281-1292. doi: 10.1111/ene.15733. Epub 2023 Feb 24. PMID 36773001
- [Derived] Siepmann T, Pinter A, Buchmann SJ, Stibal L, Arndt M, Kubasch AS, Kubasch ML, Penzlin AI, Frenz E, Zago W, Horvath T, Szatmari S Jr, Bereczki D, Takats A, Ziemssen T, Lipp A, Freeman R, Reichmann H, Barlinn K, Illigens BM. Cutaneous Autonomic Pilomotor Testing to Unveil the Role of Neuropathy Progression in Early Parkinson's Disease (CAPTURE PD): Protocol for a Multicenter Study. Front Neurol. 2017 May 26;8:212. doi: 10.3389/fneur.2017.00212. eCollection 2017. PMID 28603514
- See also: Michael J. Fox Foundation Grant Site of CAPTURE PD — https://www.michaeljfox.org/foundation/grant-detail.php?grant_id=1476